CLINICAL TRIAL: NCT02456805
Title: Efficacy of Alternate Formula Feedings in Formula Intolerant Infants
Brief Title: Alternate Formula Feedings in Formula Intolerant Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: AH23
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Gastrointestinal Tolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infant Formula 1 (Active Comparator): A standard commercial milk-based infant formula
  Interventions: Other: Infant Formula 1
- Infant Formula 2 (Experimental): A standard commercial soy-based infant formula.
  Interventions: Other: Infant Formula 2

INTERVENTIONS:
Other: Infant Formula 1 — Feed ab libitum
  Arms: Infant Formula 1
Other: Infant Formula 2 — Feed ab libitum
  Arms: Infant Formula 2

SUMMARY:
This study assessed tolerance improvement of a formula change in healthy term infants with perceived intolerance to their current milk-based formula feeding.

ELIGIBILITY:
Inclusion Criteria:

* Infants formula-fed exclusively and experiencing symptoms of cow's milk formula intolerance.
* Infants whose physicians had made a recommendation that the parents change the infant's feeding.
* Full term infants at birth with a gestational age of 37 to 42 weeks.
* Infants 2- 9 weeks of age at study entry with birth weights greater than 2500 grams.

Exclusion Criteria:

* Infants with a maternal medical history which had adverse effects on the fetus, such as diabetes, tuberculosis, perinatal infections, or substance abuse.
* Infants with evidence of cardiac, respiratory, gastrointestinal, hematological, or metabolic disease.

Ages: 2 Weeks to 9 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 1996-08; Primary Completion 1997-06 (Actual); Study Completion 1997-06 (Actual)

PRIMARY OUTCOMES:
Stool Characteristics | Change from Baseline (Study Day 1) to Study Day 15
  Parent questionnaire

SECONDARY OUTCOMES:
Formula Intake | Change from Baseline (Study Day 1) to Study Day 15
  Parent questionnaire on volume consumed
Incidence of spit up/vomiting | Change from Baseline (Study Day 1) to Study Day 15
  Parent questionnaire
Weight | Change from Baseline (Study Day 1) to Study Day 15
  Measured weight at visits

CONTACTS AND LOCATIONS:
Overall Officials: John Lasekan, MBA, Ph.D, CCRP, Study Chair — Abbott Nutrition
Locations (8):
- United States (7):
  - Arkansas Children's Hospital, Little Rock, Alaska
  - Aurora Pediatric Associates, Aurora, Colorado
  - Northlake Pediatric, Associates, Stone Mountain, Georgia
  - The Medical Associates Clinic, Dubuque, Iowa
  - Baystate Medical Center, Children's Hospital, Springfield, Massachusetts
  - Clinical Studies, Inc, Canton, Ohio
  - Richmond Pediatrics, Richmond, Virginia
- Optimum Clinical Research, Oshawa, Canada